CLINICAL TRIAL: NCT03655912
Title: Binocular Visual Therapy and Video Games for Amblyopia Treatment.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Karim Mohamed-Noriega, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OF17-00013
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Amblyopia
Keywords: Amblyopia; Binocular therapy; Videogames
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Neither the patient or the care provider will be aware of the treatment modality group the patient is in. In order to achieve that, patients in different modality groups will be evaluated in different days preventing information of group modality gossip between the patients parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patch (Active Comparator): Eye patch on the fellow eye and to near-vision activities (such as reading, drawing, etc)
  Interventions: Device: Eye patch
- Electronic Devices (Experimental): Eye patch on the fellow eye and a electronic tablet
  Interventions: Device: Electronic Tablet
- Red/Green Glasses (Experimental): Red/green glasses and a electronic tablet
  Interventions: Device: Red/green glasses

INTERVENTIONS:
Device: Red/green glasses — The use of red/green glasses and electronic devices for two hours a day during 4 months.
  Arms: Red/Green Glasses
Device: Electronic Tablet — The use of eye patch on the fellow eye and electronic tablet for 2 hours a day during 4 months.
  Arms: Electronic Devices
Device: Eye patch — The use of eye patch on the fellow eye and near vision activities for 2 hours a day during 4 months.
  Arms: Patch

SUMMARY:
Amblyopia, or lazy eye, is best defined by the American Academy of Ophthalmology as a unilateral or bilateral reduction of the best corrected visual acuity that occurs in the setting of an otherwise normal eye, or a structural abnormality involving the eye or visual pathway with reduction in visual acuity that cannot be attributed only to the effect of the structural abnormality. Which causes an abnormal visual experience early in life, with consequences such as deficiencies in the ability to perceive contrast and/or movement, visual acuity, accommodation and stereopsis. The treatment of choice consists in patching of the fellow eye 2 hours per day. The disadvantage of this treatment modality is that patients end up not complying and when treatment is interrupted, lazy eye reappears. Amblyopia was thought to be a monocular disease, now a days there are reports of cortical visual paths changes in both eyes (the fellow and amblyopia eye), believing that it might be a monocular consequence of a binocular disease. Following that statement new treatment studies have arisen, stimulating both eyes not only to improve visual acuity in the lazy eye, but to restore binocular function as well. These treatments use videogames in celular phones, computers, or tablets where the fellow eye is exposed to reduced contrast and the lazy eye is exposed to full-contrast. Although the evidence is promising, more studies are needed to establish effectivity and security of this treatment modality.

DETAILED DESCRIPTION:
The objective of this study is to determine if the binocular visual therapy with red-green glasses and the use of electronic devices is effective for amblyopia treatment in children.

Participants will be randomly assigned to one of three treatment modalities: Group A: eye patch on the fellow eye and to near-vision activities (such as reading, drawing, etc) Group B: an eye patch on the fellow eye and a electronic tablet Group C: red/green glasses and a electronic tablet

Treatment will be done buy the three groups daily during 2 consecutive hours, and will be completed for four months. Children will then suspend the therapy for 2 months, and will be reevaluated to determine lazy eye relapses . All groups will be compared to see which patients achieved greater improvement on visual acuity and depth perception.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anisometropic amblyopia, strabismic amblyopia or both
* Patients with out previous amblyopia treatment
* Patient with previous strabismus surgery or use of there best corrected visual acuity glasses for at least 1 month
* Birth at term gestational age
* Without any systemic or ophthalmic comorbidities
* Previous patients parent verbal and fiscal assessment.

Exclusion Criteria:

* Any other amblyopia diagnosis (deprivation)
* Any previous amblyopia treatment
* Any previous intraocular surgery
* Any ocular condition
* Any neurologic conditions or psychomotor development alterations
* Patients not able to cooperate for visual acuity or stereopsis evaluation

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity of the amblyopic eye | Basal
  Best corrected visual acuity of the amblyopic eye using the Snellen chart. Measurements will be converted to LogMar values for statistical analysis.
Best corrected visual acuity of the amblyopic eye | One month of treatment
  Best corrected visual acuity of the amblyopic eye using the Snellen chart. Measurements will be converted to LogMar values for statistical analysis.
Best corrected visual acuity of the amblyopic eye | Two months of treatment
  Best corrected visual acuity of the amblyopic eye using the Snellen chart. Measurements will be converted to LogMar values for statistical analysis.
Best corrected visual acuity of the amblyopic eye | Three months of treatment
  Best corrected visual acuity of the amblyopic eye using the Snellen chart. Measurements will be converted to LogMar values for statistical analysis.
Best corrected visual acuity of the amblyopic eye | Four months of treatment
  Best corrected visual acuity of the amblyopic eye using the Snellen chart. Measurements will be converted to LogMar values for statistical analysis.
Best corrected visual acuity of the amblyopic eye two months after treatment suspension to determine lazy eye relapses | Two months after treatment suspension.
  Best corrected visual acuity of the amblyopic eye using the Snellen chart. Measurements will be converted to LogMar values for statistical analysis.

SECONDARY OUTCOMES:
Stereopsis | Basal
  Stereopsis measurement by titmus test
Stereopsis | One month of treatment
  Stereopsis measurement by titmus test
Stereopsis | Two months of treatment
  Stereopsis measurement by titmus test
Stereopsis | Three months of treatment
  Stereopsis measurement by titmus test
Stereopsis | Four months of treatment
  Stereopsis measurement by titmus test
Stereopsis two months after treatment suspension to determine lazy eye relapses | Two months after treatment suspension.
  Stereopsis measurement by titmus test

CONTACTS AND LOCATIONS:
Overall Officials: Marissa L. Fernandez-de Luna, MD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Departamento de Oftalmologia, Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Tailor V, Bossi M, Bunce C, Greenwood JA, Dahlmann-Noor A. Binocular versus standard occlusion or blurring treatment for unilateral amblyopia in children aged three to eight years. Cochrane Database Syst Rev. 2015 Aug 11;2015(8):CD011347. doi: 10.1002/14651858.CD011347.pub2. PMID 26263202
- [Background] Kelly KR, Jost RM, Dao L, Beauchamp CL, Leffler JN, Birch EE. Binocular iPad Game vs Patching for Treatment of Amblyopia in Children: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):1402-1408. doi: 10.1001/jamaophthalmol.2016.4224. PMID 27832248
- [Background] Hunter D. Amblyopia: The clinician's view. Vis Neurosci. 2018 Jan;35:E011. doi: 10.1017/S0952523817000189. No abstract available. PMID 29905115
- [Background] Carlton J, Karnon J, Czoski-Murray C, Smith KJ, Marr J. The clinical effectiveness and cost-effectiveness of screening programmes for amblyopia and strabismus in children up to the age of 4-5 years: a systematic review and economic evaluation. Health Technol Assess. 2008 Jun;12(25):iii, xi-194. doi: 10.3310/hta12250. PMID 18513466
- [Background] Grant S, Melmoth DR, Morgan MJ, Finlay AL. Prehension deficits in amblyopia. Invest Ophthalmol Vis Sci. 2007 Mar;48(3):1139-48. doi: 10.1167/iovs.06-0976. PMID 17325157
- [Background] Grant S, Moseley MJ. Amblyopia and real-world visuomotor tasks. Strabismus. 2011 Sep;19(3):119-28. doi: 10.3109/09273972.2011.600423. PMID 21870915
- [Background] Hrisos S, Clarke MP, Kelly T, Henderson J, Wright CM. Unilateral visual impairment and neurodevelopmental performance in preschool children. Br J Ophthalmol. 2006 Jul;90(7):836-8. doi: 10.1136/bjo.2006.090910. Epub 2006 Mar 15. PMID 16540485
- [Background] Niechwiej-Szwedo E, Goltz HC, Chandrakumar M, Hirji Z, Wong AM. Effects of anisometropic amblyopia on visuomotor behavior, III: Temporal eye-hand coordination during reaching. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):5853-61. doi: 10.1167/iovs.11-7314. PMID 21540479
- [Background] O'Connor AR, Birch EE, Anderson S, Draper H; FSOS Research Group. The functional significance of stereopsis. Invest Ophthalmol Vis Sci. 2010 Apr;51(4):2019-23. doi: 10.1167/iovs.09-4434. Epub 2009 Nov 20. PMID 19933184
- [Background] Rahi JS, Cumberland PM, Peckham CS. Does amblyopia affect educational, health, and social outcomes? Findings from 1958 British birth cohort. BMJ. 2006 Apr 8;332(7545):820-5. doi: 10.1136/bmj.38751.597963.AE. Epub 2006 Mar 6. PMID 16520328
- [Background] Webber AL, Wood JM, Gole GA, Brown B. The effect of amblyopia on fine motor skills in children. Invest Ophthalmol Vis Sci. 2008 Feb;49(2):594-603. doi: 10.1167/iovs.07-0869. PMID 18235004
- [Background] Guo CX, Babu RJ, Black JM, Bobier WR, Lam CS, Dai S, Gao TY, Hess RF, Jenkins M, Jiang Y, Kowal L, Parag V, South J, Staffieri SE, Walker N, Wadham A, Thompson B; BRAVO study team. Binocular treatment of amblyopia using videogames (BRAVO): study protocol for a randomised controlled trial. Trials. 2016 Oct 18;17(1):504. doi: 10.1186/s13063-016-1635-3. PMID 27756405